CLINICAL TRIAL: NCT06746194
Title: The Value of 68Ga-FAPI PET/CT in the Efficacy Evaluation of Advanced Unresectable Hepatocellular Carcinoma Patients Undergoing Systemic Antitumor Therapy
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Jiajia, Deputy director, Ruijin Hospital
Other Study IDs: RuijinH 2024-541
Record Dates: First submitted 2024-12-16; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: hepatocellular carcinoma; 68Ga-FAPI; PET/CT
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients diagnosis of advanced unresectable hepatocellular carcinoma

SUMMARY:
This study aims to investigate the value of 68Ga-FAPI PET/CT in the efficacy evaluation of advanced unresectable hepatocellular carcinoma patients undergoing systemic antitumor therapy.

DETAILED DESCRIPTION:
The investigators will number all participants, create a medical record file, and record their basic information (gender, age) as well as contact information and medical history information. All participants will undergo a 68Ga-FAPI PET/CT before treatment and after 3-month treatment. The imaging response measurements will be compared with the histopathological results as gold standard.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological and clinical diagnosis of advanced unresectable hepatocellular carcinoma patients.
2. Signed and dated informed consent form.
3. Commitment to comply with research procedures and co-operation in the implementation of the full research process.
4. Aged 18-75 years old.

Exclusion Criteria:

1. Patients with serious illnesses that researchers consider unsuitable for participation in this clinical study. Such as severe heart and lung failure, severe bone marrow suppression, severe liver and kidney dysfunction, etc.
2. Intestinal perforation, complete intestinal obstruction
3. Pregnant women and women who may be pregnant, women who are breastfeeding.
4. Non-compliant person

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients and outpatients at Ruijin Hospital who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The responses to systemic antitumor therapy of advanced unresectable hepatocellular carcinoma | Within 1 week of enrollment and up to 3 months
  The tumor lesions were evaluated within one week of enrollment and at 3 months of treatment, and a comparison was made before and after. Those with improved tumor lesions were considered to have responded to the treatment, while those without improved tumor lesions were considered to have no response to the treatment.
Standardized uptake value(SUV) | Within 1 week of enrollment and after up to 3 months
  SUV of 68Ga-FAPI uptake on PET/CT images for tumor lesions

SECONDARY OUTCOMES:
Progress free survival | 3 years
  Progress free survival
Overall survival | 3 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No